CLINICAL TRIAL: NCT00685958
Title: Multicenter, Non-comparative, Open-label Study to Evaluate the Safety and Efficacy of Enoxaparin Sodium (RP54563) 20 mg Bid for 14 Days in Patients With Hip Fracture Surgery
Brief Title: Japanese Safety and Efficacy Study of Enoxaparin in Patients With Hip Fracture Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: International Clinical Development, Study Director, sanofi-aventis
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SFY6771
Record Dates: First submitted 2008-05-26; First posted 2008-05-29 (Estimated); Last update posted 2009-10-02 (Estimated); Status verified 2009-10

CONDITIONS: Hip Fractures
Keywords: Blood thinner; enoxaparin; hip fracture surgery; bleeding; thromboembolism
MeSH Terms: conditions — Hip Fractures; Hemorrhage; Thromboembolism | interventions — Enoxaparin

INTERVENTIONS:
Drug: enoxaparin (XRP4563) — 14 days of treatment

SUMMARY:
The purpose of this study is to evaluate the effects of enoxaparin on bleeding and venous blood clots in patients with hip fracture surgery.

ELIGIBILITY:
Inclusion Criteria:

* femoral neck inside or outside fracture

Exclusion Criteria:

* any major surgery on lower limbs within 3 months
* clinical signs of deep vein thrombosis
* use of non-steroidal anti-inflammatory drugs
* severe hepatic disease or renal insufficiency

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2006-07; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
bleeding events | 28 days

SECONDARY OUTCOMES:
incidence of venous thromboembolism | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (1):
- Sanofi- Aventis Administrative Office, Tokyo, Japan